CLINICAL TRIAL: NCT04077021
Title: A Phase 1, Open-label Study in Two Parts, Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of CCW702 in Patients With Metastatic, Castration Resistant Prostate Adenocarcinoma
Brief Title: First-in-human Study of CCW702 in Patients With Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBR-CCW702-3001
Record Dates: First submitted 2019-08-20; First posted 2019-09-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Castration-Resistant Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1a: Dose Escalation QOD (Experimental): CCW702 administered subcutaneously QOD, dose escalating cohorts.
  Interventions: Drug: CCW702
- Part 1b: Dose Escalation Q7D (Experimental): CCW702 administered subcutaneously Q7D, dose escalating cohorts.
  Interventions: Drug: CCW702
- Part 2: Dose Expansion (Experimental): CCW702 administered subcutaneously Q7D at RP2D.
  Interventions: Drug: CCW702

INTERVENTIONS:
Drug: CCW702 — Investigational immunotherapy for prostate cancer

SUMMARY:
CCW702 is an investigational immunotherapy for prostate cancer. This is a two-part, first-in-human study to assess the safety and tolerability of CCW702 administered subcutaneously to patients with metastatic, castration resistant prostate cancer. Part I is divided in to two subparts, in both subparts patients will receive ascending dosages of CCW702 with the goal to determine the maximum tolerated dose (MTD) of CCW702 and efficacious regimen. Part Ia will explore every other other day dosing (QOD); Part Ib will explore weekly dosing (Q7D). In part II of the study, patients will be given the recommended part/phase 2 dose (RP2D) Q7D. The study will also assess the pharmacokinetics and pharmacodynamics of CCW702.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years of age at time of informed consent
* For Part 1 and Part 2: men with metastatic castration resistant prostate cancer (mCRPC) with histologically or cytologically confirmed adenocarcinoma of the prostate as defined by one or more of the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria
* Patients with treated brain metastasis or LMD are eligible if brain imaging shows no evidence of progression
* Must have prostate-specific antigen (PSA) and/or radiographic progression on AT LEAST One novel androgen receptor (AR)-targeted therapy (abiraterone acetate, enzalutamide).
* Eastern Cooperative Oncology Group performance status of 0-1
* Adequate liver function
* Adequate hematopoietic function
* Testosterone level ≤ 50 ng/mL (or 1.73 nmol/L)
* Patient has a life expectancy of greater than 12 weeks

Exclusion Criteria:

* Patients whose tumors solely exhibit neuroendocrine differentiation or small cell features by histopathology
* Patients with new or progressive brain metastasis or Leptomeningeal Disease (LMD)
* Patients with a history of clinically significant cardiovascular disease such as symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, history of stroke or myocardial infarction within 6 months of enrollment
* Patients with peripheral neuropathy CTCAE Grade >/= 2
* Patients with a known history of hypersensitivity, allergy or intolerance to CCW702 or its excipients
* Patients with untreated or imminent spinal cord compression

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Part 1a and 1b: Assess the safety and tolerability of CCW702, including incidence of dose limiting toxicities | up to day 28
  Frequency, severity, duration of treatment-emergent and treatment-related adverse events per CTCAE v5.0
Part 1a and 1b: Select recommended phase/part 2 dose | up to 2 years
  Review of safety and tolerability data (adverse events, dosing) based on CTCAE v5 of all Part 1 subjects/cohorts
Part 2: to assess clinical efficacy at the RP2D | up to 2 years
  Responses will be measured using prostate cancer working group 3 (PCWG3) criteria

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California at San Diego, San Diego, California
  - Johns Hopkins University - Sydney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim CH, Axup JY, Lawson BR, Yun H, Tardif V, Choi SH, Zhou Q, Dubrovska A, Biroc SL, Marsden R, Pinstaff J, Smider VV, Schultz PG. Bispecific small molecule-antibody conjugate targeting prostate cancer. Proc Natl Acad Sci U S A. 2013 Oct 29;110(44):17796-801. doi: 10.1073/pnas.1316026110. Epub 2013 Oct 14. PMID 24127589
- [Derived] Lee SC, Ma JSY, Kim MS, Laborda E, Choi SH, Hampton EN, Yun H, Nunez V, Muldong MT, Wu CN, Ma W, Kulidjian AA, Kane CJ, Klyushnichenko V, Woods AK, Joseph SB, Petrassi M, Wisler J, Li J, Jamieson CAM, Schultz PG, Kim CH, Young TS. A PSMA-targeted bispecific antibody for prostate cancer driven by a small-molecule targeting ligand. Sci Adv. 2021 Aug 11;7(33):eabi8193. doi: 10.1126/sciadv.abi8193. Print 2021 Aug. PMID 34380625